CLINICAL TRIAL: NCT02830997
Title: A Comparison of Surgical Technologies for Accuracy of Prosthesis Placement and Ease of Surgeon Use in Total Knee Arthroplasty
Brief Title: Total Knee Arthroplasty Guidance Systems Study
Status: Completed | Type: Observational
Sponsor: Ormonde M. Mahoney, MD (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor-Investigator, Ormonde M. Mahoney, MD, Principal Investigator, Athens Orthopedic Clinic, P.A.
Organization: Athens Orthopedic Clinic, P.A. (Other)
Other Study IDs: AOC-OM-St-2015-026
Record Dates: First submitted 2016-07-09; First posted 2016-07-13 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Conventional guidance: The conventional guidance will undergo TKA surgery with use of the Investigator's usual precision guided technique based on conventional instrumentation (mechanical and simple computer-assisted guidance techniques). For participants of the conventional guidance arm, the Investigator will employ the established technique he currently employs for all routine TKA procedures and would employ if the patient were not a participant in the study.
- Stereotactic guidance: The stereotactic guidance group will undergo their TKA surgery with use of a stereotactic guidance system.
  Interventions: Device: Stereotactic guidance system

INTERVENTIONS:
Device: Stereotactic guidance system
  Other Names: Stryker robotic arm system (Mako)
  Groups: Stereotactic guidance

SUMMARY:
In total knee replacement operations, the surgeon uses techniques and instruments to guide the operation and ensure that all parts of the prosthesis (the artificial knee surfaces) are placed into the correct position. There are many techniques a surgeon can use to achieve accuracy in the operation. This study will compare the Principal Investigator's present precision-guided technique and instrumentation methods with a newly developed technique that uses a computer-based stereotactic guidance system. The purposes of the study are: 1.) to learn whether the use of the different guidance systems results in differences of accuracy of the placement of the prosthesis; 2.) to compare the length of time it takes an experienced joint replacement specialist to complete the operation using the different guidance systems; 3.) to learn whether there are advantages of either system in terms of the function and recovery of patients over the first year after surgery; and, 4.) to provide the manufacturer of the stereotactic guidance system with feedback on the technical ease of use and workflow ease of the system which may be used for training and education purposes and/or for planning further refinements to the system. The study will enroll up to 150 patients from Athens Orthopedic Clinic over 2 to 3 years.

DETAILED DESCRIPTION:
The open-label study aims to enroll up to 75 participants into the conventional guidance arm followed by 75 participants into the stereotactic guidance arm, in sequence.

Detailed observational data will be collected during the surgical procedures, and participating patients will be evaluated at prescribed intervals (pre-operatively, and 2,4,6, and 12 months post-operatively) using survey instruments, clinical indicators, and routine radiologic outcomes. Radiologic outcomes will be assessed using standard x-rays that are obtained in the course of normal care for all patients who undergo total knee arthroplasty (TKA). A subset of the first 30 patients enrolled into each treatment arm will, in addition, be asked to voluntarily undergo a computed tomography (CT) scan of the lower extremity (hip, knee, and ankle joints) 8-12 weeks after surgery to measure 3-dimensional accuracy of prosthesis placement and limb alignment.

Data collection will include:

1. Demographic and background information (age, sex, height, weight, social (occupation/employment), major comorbidity (broadly classified), smoking)
2. Patient reported outcome measures (Veteran's Rand 12-item Health Survey; 2011 Knee Society Score)
3. Physical Examination (knee range of motion, knee stability)
4. Details of the surgical operation
5. Operating room workflow details, including skin-to-skin surgical time
6. Post-operative disposition
7. Radiologic outcomes

   1. Routine pre- and post-operative radiographs will be reviewed for limb alignment and evidence of prosthesis fixation
   2. Post-operative CT scans (hip, knee, ankle) will be used to evaluate accuracy of placement of the TKA prosthesis (femoral and tibial components) and accuracy of limb alignment in the coronal, sagittal, and axial planes. The values measured from the post-operative CT scan will be compared to those of the final intra-operative plan; lack of difference between the two will constitute 'accuracy'.
8. Adverse events
9. Patients may optionally participate in an additional clinical follow-up visit at 2 years post-operatively, which will include the patient reported outcome measures, physical, examination, and radiographic examination.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo unilateral primary total knee arthroplasty performed by the Principal Investigator at St. Mary's Hospital
2. Use of Triathlon® CR Total Knee System is indicated
3. Spinal anesthetic is planned
4. Age 45 years or greater
5. Body mass index (BMI) ≤ 40 kg/m2
6. Patient is willing and able to undergo postoperative follow-up requirements and self evaluations
7. Patient gives valid informed consent and signs the approved Informed Consent and Protected Health Information Use Authorization forms

Exclusion Criteria:

1. Age < 45 years
2. BMI > 40 kg/m2
3. General anesthetic is planned
4. Patient scheduled for bilateral total knee arthroplasty, or plans to undergo arthroplasty of another lower extremity joint within one year
5. Prior high tibial osteotomy or previous reconstruction to the affected knee including partial arthroplasty
6. Neuromuscular disorders, muscular atrophy, or vascular deficiency in the affected limb
7. Patient is skeletally immature
8. Active infection or suspected infection in or about the joint
9. Bone stock that is inadequate to support fixation of the prosthesis
10. Collateral ligament insufficiency
11. Blood supply limitations, refusal to receive blood transfusion (e.g., religious objection), or medical condition that predisposes patient to increased risk of blood loss (e.g., hemophilia)
12. Patient is non-ambulatory
13. Female patient is pregnant or lactating
14. Patient is incarcerated
15. Patient is critically ill or medically frail
16. Patient with mental or neurological conditions who may be incapable of following instructions
17. Previous history of radiation therapy, or other significant lifetime radiation exposure or contraindication to voluntary medical radiation exposure
18. Has previously participated in or was previously invited to participate in this study during surgery of the contralateral knee, or was previously invited to participate in the opposite treatment arm during surgery of the same knee.
19. Cannot or does not give valid informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source of participants for this study will be the pool of patients who have already elected to undergo TKA surgery under the Principal Investigator's care and have requested a surgery date with the scheduling nurse. The study population will consist of men and women aged 45 years and older selected from this source population at the discretion of the investigator who meet the eligibility criteria and voluntarily enroll in the study. There will be no solicitation of potential participants from the community or seeking of referrals for the purposes of recruitment into this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of total knee arthroplasty component placement in the coronal, axial, and sagittal planes measured by computed tomography scan | 2 months post-operatively
  Difference of coronal alignment between pre-operative plan and resultant alignment measured by post-operative CT scan

SECONDARY OUTCOMES:
Skin-to-skin surgical time in minutes | measured during the surgical operation
  Skin-to-skin surgical time in minutes
Patient reported physical function measured by 2011 Knee Society Scoring System | 2, 4, 6, and 12 months post-operatively
  Patient reported physical function measured by 2011 Knee Society Scoring System
Patient reported health related quality of life measured by the Veteran's Rand 12-item Health Survey | 2, 4, 6, and 12 months post-operatively
  Patient reported health related quality of life measured by the Veteran's Rand 12-item Health Survey
Patient reported satisfaction measured by 2011 Knee Society Scoring System | 2,4,6, and 12 months post-operatively
  Patient reported satisfaction measured by 2011 Knee Society Scoring System

CONTACTS AND LOCATIONS:
Overall Officials: Ormonde M Mahoney, MD, Principal Investigator — Athens Orthopedic Clinic, P.A.; Tracy L Kinsey, MSPH, Study Director — Athens Orthopedic Clinic, P.A.
Locations (1):
- Athens Orthopedic Clinic, P.A., Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No